CLINICAL TRIAL: NCT00006518
Title: Collection of Blood, Bone Marrow, Tumor, or Tissue Samples From Patients With HIV Infection, KSHV Infection, Viral-Related Pre-Malignant Lesions, and/or Cancer
Brief Title: Specimen Collections From Participants With HIV Infection, KSHV Infection, Viral-Related Pre-malignant Lesions and Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010038; 01-C-0038; NCT00898651 (obsolete NCT alias)
Record Dates: First submitted 2000-11-22; First posted 2000-11-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: HIV; Kaposi's Sarcoma; Lymphomas; Multicentric Castleman's Disease; Primary Effusion Lymphoma
Keywords: Tumor; Viruses; HIV; KSHV; AIDS; Natural History
MeSH Terms: conditions — Sarcoma, Kaposi; Lymphoma; Multi-centric Castleman's Disease; Lymphoma, Primary Effusion; Neoplasms; Virus Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Participants with HIV infection, KSHV infection, or with cancer

SUMMARY:
BACKGROUND:

* A number of important scientific advances can be made through the study of blood, bone marrow, tumor, or other tissue samples from patients with HIV infection, infection with Kaposi s sarcoma associated herpesvirus (KSHV), infection with other oncogenic viruses, or cancer.
* This protocol provides a mechanism to affect a variety of such studies.

OBJECTIVES:

-Acquisition of serum, circulating cells, bone marrow, and tumor or normal tissue samples from participants with HIV infection, KSHV infection, or with cancer.

ELIGIBILITY:

-Eligibility criteria include age 18 years or older and at least one of the following: Exposure risk to HIV, KSHV, or HPV; HIV seropositive; KSHV seropositive; EBV seropositive; HTLV-1 seropositive; malignancy, Castleman s disease, or skin lesions with appearance of Kaposi s sarcoma; or cervical or anal intraepithelial lesion.

DESIGN:

* Up to 999 subjects will be enrolled in this study.
* Blood samples may be collected at the initial visit, and at follow-up visits.
* Other fluids/excretions may be collected (such as urine, saliva, semen, and stool).
* Tumor samples may be obtained by fine needle aspirate, by removal of pleural or peritoneal fluid, by skin punch biopsy, or by excisional biopsy, providing the tumor is accessible with minimal risk to the participants.
* Specific risks will be described in a separate consent to be obtained at the time of the biopsy.
* Samples will be studied in the HIV and AIDS Malignancy Branch, CCR, NCI; laboratories in NCI-Frederick; or those of collaborating investigators.

DETAILED DESCRIPTION:
BACKGROUND:

* A number of important scientific advances can be made through the study of blood, bone marrow, tumor, or other tissue samples from patients with HIV infection, infection with Kaposi s sarcoma associated herpesvirus (KSHV), infection with other oncogenic viruses, or cancer.
* This protocol provides a mechanism to affect a variety of such studies.

OBJECTIVES:

-Acquisition of serum, circulating cells, bone marrow, and tumor or normal tissue samples from participants with HIV infection, KSHV infection, or with cancer.

ELIGIBILITY:

-Eligibility criteria include age 18 years or older and at least one of the following: Exposure risk to HIV, KSHV, or HPV; HIV seropositive; KSHV seropositive; EBV seropositive; HTLV-1 seropositive; malignancy, Castleman s disease, or skin lesions with appearance of Kaposi s sarcoma (KS); or cervical or anal intraepithelial lesion.

DESIGN:

* Up to 999 participants will be provide samples in this study.
* Blood samples may be collected at the initial visit, and at follow-up visits.
* Other fluids/excretions may be collected (such as urine, saliva, semen, and stool).
* Tumor samples may be obtained by fine needle aspirate, by removal of pleural or peritoneal fluid, by skin punch biopsy, or by excisional biopsy, providing the tumor is accessible with minimal risk to the participants.
* Specific risks will be described in a separate consent to be obtained at the time of the biopsy.
* Samples will be studied in the HIV and AIDS Malignancy Branch, CCR, NCI; laboratories in NCI-Frederick; or those of collaborating investigators.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years or older.
* ECOG performance status less than or equal to 3

At least one of the following:

* Exposure risk to HIV, KSHV, or HPV
* HIV seropositive
* KSHV seropositive
* EBV seropositive
* HTLV-1 seropositive

NOTE: infection with HIV, KSHV, EBV, and HTLV-1 are life-long, so if participants have previously been seropositive or have had a disease associated with KSHV (KS, primary effusion lymphoma [PEL], or KSHV-multicentric Castleman s disease [MCD]), this is sufficient to meet this criterion for eligibility.

* Malignancy, MCD, or skin lesions with appearance of KS
* Cervical or anal intraepithelial lesion
* Ability of participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 1029 (Estimated)
Dates: Start 2000-12-06 (Actual)

PRIMARY OUTCOMES:
Acquisition of serum, circulating cells, bone marrow, and tumor or normal tissue samples from participants with HIV infection, KSHV infection, or with cancer. | Ongoing
  Proportion of participants that have contributed serum, circulating cells, bone marrow, and tumor or normal tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Davis DA, Dorsey K, Wingfield PT, Stahl SJ, Kaufman J, Fales HM, Levine RL. Regulation of HIV-1 protease activity through cysteine modification. Biochemistry. 1996 Feb 20;35(7):2482-8. doi: 10.1021/bi951525k. PMID 8652592
- [Background] Davis DA, Newcomb FM, Moskovitz J, Wingfield PT, Stahl SJ, Kaufman J, Fales HM, Levine RL, Yarchoan R. HIV-2 protease is inactivated after oxidation at the dimer interface and activity can be partly restored with methionine sulphoxide reductase. Biochem J. 2000 Mar 1;346 Pt 2(Pt 2):305-11. PMID 10677347
- [Background] Pinto LA, Berzofsky JA, Fowke KR, Little RF, Merced-Galindez F, Humphrey R, Ahlers J, Dunlop N, Cohen RB, Steinberg SM, Nara P, Shearer GM, Yarchoan R. HIV-specific immunity following immunization with HIV synthetic envelope peptides in asymptomatic HIV-infected patients. AIDS. 1999 Oct 22;13(15):2003-12. doi: 10.1097/00002030-199910220-00002. PMID 10546852
- [Derived] Lage SL, Ramaswami R, Rocco JM, Rupert A, Davis DA, Lurain K, Manion M, Whitby D, Yarchoan R, Sereti I. Inflammasome activation in patients with Kaposi sarcoma herpesvirus-associated diseases. Blood. 2024 Oct 3;144(14):1496-1507. doi: 10.1182/blood.2024024144. PMID 38941593
- [Derived] Ramaswami R, Tagawa T, Mahesh G, Serquina A, Koparde V, Lurain K, Dremel S, Li X, Mungale A, Beran A, Ohler ZW, Bassel L, Warner A, Mangusan R, Widell A, Ekwede I, Krug LT, Uldrick TS, Yarchoan R, Ziegelbauer JM. Transcriptional landscape of Kaposi sarcoma tumors identifies unique immunologic signatures and key determinants of angiogenesis. J Transl Med. 2023 Sep 22;21(1):653. doi: 10.1186/s12967-023-04517-5. PMID 37740179
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-C-0038.html